CLINICAL TRIAL: NCT07340268
Title: The Effects of Transcranial Current Stimulation on Insomnia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zan Wang (Other)
Responsible Party: Sponsor-Investigator, Zan Wang, Sleep Center Director, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCS-V01
Record Dates: First submitted 2026-01-04; First posted 2026-01-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Insomnia, Psychophysiological
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active transcranial current stimulation (Active Comparator): 14 daily 20-min, 1.1-mA sessions of active or sham transcranial current stimulation, at the beginning and end of treatment, there is a 30 second period of current fading in and out
  Interventions: Device: transcranial current stimulation
- sham transcranial current stimulation (Sham Comparator): only wore the device and had no stimulation
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: transcranial current stimulation — consecutive daily 20-min, 1.1-mA sessions
  Arms: active transcranial current stimulation
Device: Sham stimulation — only wore the device and had no stimulation
  Arms: sham transcranial current stimulation

SUMMARY:
Effect of transcranial current stimulation on insomnia disorder

DETAILED DESCRIPTION:
Insomnia disorder represents a prevalent clinical challenge, transcranial current stimulation has emerged as a promising noninvasive therapeutic approach; however, its specific effects on neurophysiological mechanisms underlying sleep-related brain structure and functional change, and neurobiological change remain unclear.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of insomnia disorder
* Cooperate to complete the questionnaire surveys

Exclusion Criteria:

* Presence of mental disorders
* Current use of central nervous system stimulants
* Use of analgesics,sedatives or hypnotic medications, theophylline preparations, steroid medications
* Alcohol abuse or regular alcohol consumption
* Diagnosis of other sleep disorders, including obstructive sleep apnea, rapid eye movement sleep behavior disorder, or restless legs syndrome
* Sleep disorders secondary to organic diseases, such as epilepsy, diabetes, or renal failure
* Shift work or irregular work schedules that disrupt normal circadian rhythms
* Use of medications affecting central nervous system function within the past one month
* Recent sleep-related confounding behaviors within the past two weeks, including staying up late, alcohol consumption, or smoking
* Presence of organic brain lesions on head MRI and contraindications to MRI examination

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-18 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in global blood-oxygen-level-dependent (gBOLD) signal amplitude | 2 weeks and 3 months
  The amplitude of the global blood-oxygen-level-dependent (gBOLD) signal was derived from resting-state functional MRI and reflects the overall magnitude of spontaneous brain activity. Unit of Measure: Z-score
Change in resting-state functional connectivity strength | 2 weeks and 3 months
  Resting-state functional connectivity strength was calculated as the correlation coefficient between predefined brain regions based on functional magnetic resonance imaging data.
Change in amplitude of low-frequency fluctuations | 2 weeks and 3 months
  Amplitude of low-frequency fluctuations was calculated from resting-state fMRI to quantify spontaneous neural activity.
Change in regional homogeneity | 2 weeks and 3 months
  Regional homogeneity was used to assess the synchronization of local spontaneous brain activity
Change in phase difference of dynamic cerebral autoregulation | 2 weeks and 3 months
  Dynamic cerebral autoregulation was assessed using the phase difference between cerebral blood flow velocity and arterial blood pressure fluctuations. Larger phase differences indicate better autoregulatory function.
Change in gain of dynamic cerebral autoregulation | 2 weeks and 3 months
  Gain represents the magnitude of cerebral blood flow velocity changes in response to blood pressure fluctuations, with lower gain values indicating more effective autoregulation.

SECONDARY OUTCOMES:
the score of Insomnia Severity Index scale | 2 weeks and 3 months
  The total score ranges from 0 to 28, and a higher score indicates higher levels of insomnia severity. A score of 8 or greater is the cut point for clinically possible insomnia
the score of 14-item Hamilton anxiety rating scale | 2 weeks and 3 months
  The total score ranges from 0 to 56, and a higher score indicates higher levels of anxiety symptoms. A score of 7 or greater is the cut point for clinically possible anxiety
the score of 17-item Hamilton depression rating scale | 2 weeks and 3 months
  tThe total score ranges from 0 to 52, and a higher score indicates higher levels of depression symptoms. A score of 7 or greater is the cut point for clinically possible depression symptom
Change in plasma corticotropin-releasing factor (CRF) level | 2 weeks and 3 months
  Plasma corticotropin-releasing factor (CRF) concentration was measured as a biomarker of hypothalamic-pituitary-adrenal (HPA) axis activity. Higher levels indicate increased neuroendocrine stress response. Unit of Measure: pg/mL
Change in plasma cortisol level | 2 weeks and 3 months
  Plasma cortisol concentration was assessed as an indicator of hypothalamic-pituitary-adrenal (HPA) axis function. Higher levels reflect increased physiological stress response. Unit of Measure: μg/dL
Change in serum interleukin-6 level | 2 weeks and 3 months
  Serum interleukin-6 concentration was measured as a marker of systemic inflammation. Higher levels indicate greater inflammatory activity. Unit of Measure: pg/mL
Change in serum brain-derived neurotrophic factor level | 2 weeks and 3 months
  Serum brain-derived neurotrophic factor concentration was measured as a biomarker associated with neuroplasticity and neuronal function. Higher levels indicate enhanced neurotrophic activity. Unit of Measure: pg/mL
Change in total sleep time (TST) measured by polysomnography | 2 weeks and 3 months
Change in sleep onset latency (SOL) measured by polysomnography | 2 weeks and 3 months
Change in wake after sleep onset (WASO) measured by polysomnography | 2 weeks and 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of Jilin University, Ch’ang-ch’un, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided